CLINICAL TRIAL: NCT02165670
Title: BioMatrix NeoFlex Post Marketing Surveillance in Validate (the BASIC VALIDATE) Registry)
Brief Title: BASIC VALIDATE Coronary Stent Registry
Status: Withdrawn | Type: Observational
Why Stopped: After critique raised by peers there was a risk that the study could be interpreted as a marketing tool for a specific product more than a scientific study.
Sponsor: Region Örebro County (Other)
Collaborators: Biosensors International (Other)
Responsible Party: Principal Investigator, Ole Frobert, MD, PhD, Adjunct Professor, MD, PhD, Region Örebro County
Other Study IDs: BASIC VALIDATE; Prospective registry
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Myocardial Infacrtion; Unstable Angina Pectoris; Stable Angina Pectoris
Keywords: Ischemic heart disesase; Myocardial infarction; Angina pectoris
MeSH Terms: conditions — Angina, Unstable; Angina, Stable; Myocardial Infarction; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ischemic heart disease: Patients undergoing percutaneous coronary intervention (PCI)
  Interventions: Device: Coronary stenting with CE-marked stent

INTERVENTIONS:
Device: Coronary stenting with CE-marked stent
  Other Names: BioMatrix Flex™ stent (Biosensors International)

SUMMARY:
BASIC VALIDATE is a coronary stent registry to obtain clinical follow-up information from 2000 patients treated with CE-marked stent (BioMatrix Flex™, Biosensors International) with follow-up of endpoints via the Swedish angiography and angioplasty registry (SCAAR - part of the national SWEDEHEART registry).

DETAILED DESCRIPTION:
Purpose of the study The purpose of this registry is to capture clinical data of the BioMatrix NeoFlex™ stent (an improved version of the delivery system of the Biolimus A9™-eluting BioMatrix Flex stent) in relation to safety and effectiveness in the VALIDATE SWEDEHEART trial and in a group of patients not taking part in VALIDATE SWEDEHEART in addition to a group of patients with stable angina pectoris.

Clinical relevance The European Union has a focus on and encourages the conductance of post marketing surveillance studies of medical devices 3. This focus should be seen in the light of limitations to clinical data available in the pre-market phase owing to duration of pre-market clinical investigations, the number of subjects and investigators involved in an investigation, the relative heterogeneity of subjects and investigators and the controlled setting of a clinical investigation versus the full range of clinical conditions encountered in general medical practice. The extent of the data that can be gathered in the pre-market phase does not necessarily enable detection of rare complications or problems that only become apparent after widespread or long term use of the device. Because the study device (BioMatrix NeoFlex™) is a CE-marked updated version of the BioMatrix Flex stent it is important to document that the assumed improvements in delivery design also reflect improvements in a clinical setting.

Patients and methods

Patients A total of 6000 patients will be included in the VALIDATE SWEDEHEART trial. 3000 STEMI and 3000 NSTEMI. The ambition is that approximately 1000 of these patients are also included in the BASIC VALIDATE stent registry. In addition, and in order to achieve post-market information from the entire spectrum of PCI, another 1000 patients with stable angina pectoris, STEMI or NSTEMI will be included in the registry at VALIDATE SWEDEHEART centers but unrelated to the VALIDATE SWEDEHEART trial.

Treatment strategy During the index procedure, only BioMatrix NeoFlex™ stents will be implanted. The investigator will choose the appropriate length and diameter of the stents to be implanted by visual estimate. The choice of the length of the stent should ensure complete coverage of the lesion. In case of insufficient stent expansion, post-dilatation is highly recommended. In the event that a staged procedure is expected or planned it is recommended NOT to include the patient in the BASIC VALIDATE registry because the nature of follow-up of patients (registry only) means that staged procedures will be classified as events ("repeat" revascularizations).

After the index PCI, lifelong acetylsalicylic acid in a dose of 75-160 mg per day will be prescribed. Duration and choice of post-PCI P2Y12 inhibition is left to the discretion of the treating physician.

Endpoints Primary endpoint A composite of time to death, myocardial infarction, stent thrombosis or repeat revascularization at 12 months.

Secondary endpoints

* Time to death at 1, 3 and 5 years.
* Time to myocardial infarction at 1, 3 and 5 years.
* Time to stent thrombosis at 1, 3 and 5 years.
* Time to repeat revascularization at 1, 3 and 5 years.
* Analysis of the primary endpoint in the NSTEMI and STEMI groups separately.

All endpoint results will be compared to matched populations of patients treated with drug-eluting coronary stents as documented in the SCAAR/SWEDEHEART registries.

ELIGIBILITY:
Inclusion Criteria

* Patients with a diagnosis of NSTEMI as judged by the physician in accordance with current guideline definitions (positive troponin).
* Patients with a diagnosis of STEMI as defined by chest pain suggestive for myocardial ischemia for at least 30 minutes before hospital admission, time from onset of symptoms of less than 24 hours, and an ECG with new ST-segment elevation in two or more contiguous leads of ≥0.2 mV in leads V2-V3 and/or ≥0.1 mV in other leads or a probable new-onset left bundle branch block.
* Patients with stable coronary artery disease
* PCI of culprit lesion is intended.
* Age above 18 years

Exclusion Criteria:

* Previous participation in the BASIC VALIDATE registry
* Known terminal disease with life expectancy less than one year.
* Patients with known ongoing bleeding
* Patients with uncontrolled hypertension in the opinion of the investigator
* Patients with known subacute bacterial endocarditis
* Patients with known severe renal (GFR < 30 ml/min) and /or liver dysfunctions
* Patients with known thrombocytopenia or thrombocyte function defects

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic heart disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Death, MI, Stent Thrombosis, Revascularization | 1 year
  A composite of time to death, myocardial infarction, stent thrombosis or repeat revascularization at 12 months.

SECONDARY OUTCOMES:
Long time Death, AMI, Stent Thrombosis, Revascularization | 5 years
  Time to death at 1, 3 and 5 years, time to myocardial infarction at 1, 3 and 5 years, time to stent thrombosis at 1, 3 and 5 years, time to repeat revascularization at 1, 3 and 5 years.